CLINICAL TRIAL: NCT00133861
Title: Botulinum Toxin Efficiency on Spasticity of Rectus Femoris and Semitendinosus Muscles as Functional Agonist and Antagonist Muscles. Assessment of Efficiency of Botulinum Toxin on Spasticity in Agonist and Antagonist Muscles Using Clinical Assessment and Gait Analysis in Cerebral Palsy Children: Rectus Femoris and Semitendinosus
Brief Title: Botulinum Toxin Efficiency on Spasticity of Rectus Femoris and Semitendinosus Muscles as Functional Agonist and Antagonist Muscles
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004.351
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy children; Botulinum toxin
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins

INTERVENTIONS:
Drug: Botulinum toxin

SUMMARY:
The aim of the study is to confirm the functional improvement obtained through treatment of spasticity on 2 agonist and antagonist muscles. The hypothesis is that treatment of both muscles gives a better and longer functional improvement than treatment of only one muscle. The target muscles are the rectus femoris and semitendinosus and the treatment is botulinum toxin. Clinical assessment (passive range of motion of the lower limbs, spasticity level, functional scales and subjective feeling) and gait analysis data (kinematics and kinetics data) are collected. Evaluations take place before treatment, 2 months and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 7 to 17 years old
* Cerebral palsy children with walking ability (even with crutch or knee-walker) allowing gait analysis.
* Patients with functional status allowing the use of botulinum toxin on target muscles.

Exclusion Criteria:

* Patients under 7 years old
* Patients up to 17 years old
* Patients in whom botulinum toxin is contra-indicated
* Patients who received botulinum toxin within a 6 month period before the beginning of the study

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Estimated)
Dates: Start 2005-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of the passive range of motion of the lower limbs

SECONDARY OUTCOMES:
Evaluation of the spasticity using Tardieu Scale, Ashworth Scale and Ely test
Evaluation of functional outcome using Gross Motor Function Measure and Gillette Functional Assessment, subjective evaluation, physiological cost index

CONTACTS AND LOCATIONS:
Overall Officials: Bruno DOHIN, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot - Pavillon T bis, Lyon, France

REFERENCES:
- [Result] Dohin B, Garin C, Vanhems P, Kohler R. [Botulinum toxin for postoperative care after limb surgery in cerebral palsy children]. Rev Chir Orthop Reparatrice Appar Mot. 2007 Nov;93(7):674-81. doi: 10.1016/s0035-1040(07)73252-x. French. PMID 18065878